CLINICAL TRIAL: NCT04168034
Title: The iParent2Parent Program: Peer Mentoring for Parents of Children With Juvenile Idiopathic Arthritis
Brief Title: iParent2Parent Program for Parents of Children With Juvenile Idiopathic Arthritis
Acronym: iPa2PaJIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Sara Ahola Kohut, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000061063
Record Dates: First submitted 2019-10-18; First posted 2019-11-19 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: JIA

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: iParent2Parent Mentorship (Experimental): 10 sessions of 20-30 minute Skype video calls conducted over 2 to 3 months
  Interventions: Behavioral: iParent2Parent Program
- Waitlist Control Group (Active Comparator): The control group will receive standard care but without the iParent2Parent program
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: iParent2Parent Program — In addition to standard care, parents in the experimental group will receive the iParent2Parent program. The iParent2Parent program is a tailored peer mentorship program that provides modeling and reinforcement by peers (trained parents of children with JIA) to parents of children diagnosed with JIA.
  Arms: Experimental: iParent2Parent Mentorship
Behavioral: Waitlist Control — The control group will receive standard care but without the iParent2Parent program
  Arms: Waitlist Control Group

SUMMARY:
The iParent2Parent program matches parents of children living with arthritis with a trained parent mentor who will provide parents of children newly diagnosed with arthritis: practical coping advice and social support through shared lived experiences. This study will compare two groups of parents: those who are in the iParent2Parent program and those in the control group (no mentor).

DETAILED DESCRIPTION:
Parents/primary caregiver of children with JIA are an often overlooked but essential member of their child's health care team. They are responsible for managing their child's treatment program, and act as advocates for their child to support positive adaptation to JIA and to learn self-management skills for the disease. This is in the context of managing the financial, logistical, emotional, and social demands of parenting in general. Within pediatric tertiary care centres, peer-support programs for parents of children with JIA are often limited or difficult to access. The iParent2Parent Program aims to fill this gap in services by offering a program of trained parent peer mentors who can provide practical coping advice, foster adaptive problem solving, and provide social support via shared lived experience.

ELIGIBILITY:
Inclusion Criteria:

* English speaking caregiver of a child diagnosed with JIA according to ILAR criteria prior to their 18th birthday
* Access to computer capable of using free Skype software

Exclusion Criteria:

* Significant cognitive impairment or major co-morbid illness of parent that impeded ability to engage in program (e.g.; psychosis, active suicidal ideation, cognitive delays that would impact ability to participate and complete questionnaires.)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Trial feasibility of iParent2Parent program | At study completion; an average of 2 years
  Criteria for feasibility are based on studies previously conducted by our group and will be: accrual rate of >70 percent, attrition rate of <15percent, technical difficulties reported by <10 percent of parents and mentors, adherence rate of >80 percent, <5 percent missed responses on outcome measures and high acceptability (based on qualitative analyses). Data related to the primary outcome will be recorded on investigator-developed forms.

SECONDARY OUTCOMES:
PROMIS Adult Profile 25 | baseline; up to 12 weeks after baseline, 6 months post program
  29 item collection of short forms from 7 health domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance and ability to participate in social roles and activities. The scale is scored from 1 to 5. The higher the score the worse the outcome
Short form version of the PROMIS | baseline; up to 12 weeks after baseline, 6 months post program
  Short form version of the PROMIS battery for Social Isolation; Informational support; and Emotional support. The scale is scored from 1 to 5. The higher the score the better the outcome (emotional and informational support). The higher the score the worse the outcome for social isolation)
Coping Health Inventory for Parents | baseline; up to 12 weeks after baseline, 6 months post program
  45-item measure of a parent's response to managing demands when a child has a serious or chronic medical condition. The lower the score, the worse the outcome. Minimum value 0 and maximum value 3.
Parental Stress Scale | baseline; up to 12 weeks after baseline, 6 months post program
  Attempts to measure the levels of stress experienced by parents. The scale is scored from 1 to 5. The lower the score the lower the level of stress and the higher the score the higher the level of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ahola Kohut, PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - The IWK Health Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT04168034/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT04168034/SAP_001.pdf